CLINICAL TRIAL: NCT04822649
Title: Differences in Cardiopulmonary Exercise Capacity According to Coronary Microvascular Dysfunction and Body Composition in Patients With Suspected Heart Failure With Preserved Ejection Fraction
Brief Title: Exercise Capacity According to Coronary Microvascular Dysfunction and Body Composition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Seong-Mi Park, M.D. Ph.D., Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020AN0030
Record Dates: First submitted 2021-03-18; First posted 2021-03-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: body composition, CPET, CFR, coronary microvascular dysfunction (CMD), frailty, HFpEF
MeSH Terms: conditions — Frailty | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Patients with chest pain or ischemic symptoms with non-obstructive coronary artery disease (<50% stenosis) in coronary angiography and preserved ejection fraction (>50%) in echocardiography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heart failure with preserved ejection fraction (Other): Adenosine stress echocardiography, body composition, and cardiopulmonary exercise test will be done in all of the enrolled patients. Left ventricular end-diastolic pressure will be assessed during coronary angiography.
  Interventions: Diagnostic Test: Adenosine stress echocardiography with the evaluation of coronary artery blood flow

INTERVENTIONS:
Diagnostic Test: Adenosine stress echocardiography with the evaluation of coronary artery blood flow — The color Doppler flow of distal left anterior descending artery will be examined from the modified apical four-chamber view in the anterior interventricular groove.
  In regard to body composition analysis, Using InBody S10, impedance is measured in 6 frequency bands (1 kilohertz (kHz), 5 kHz, 50 kHz, 250 kHz, 500 kHz, 1000 kHz) for each of 5 parts (right plate, left arm, torso, right leg, left leg). Reactance is measured in 3 frequency bands (5 kHz, 50 kHz, 250 kHz for each of 5 parts (right arm, left arm, torso, right leg, left leg).
  By treadmill exercise test with modified Bruce protocol or bicycle ergometer for patients with orthopedic problems, maximal oxygen consumption (VO2 max) will be measured using the exhalation gas analysis.
  Other Names: Body composition analysis; Cardiopulmonary exercise test

SUMMARY:
The correlation of coronary microvascular function and body composition with cardiopulmonary exercise capacity will be assessed in patients with heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
We will select the patients with chest pain or ischemic symptoms with non-obstructive coronary artery disease (<50% stenosis) in coronary angiography and preserved ejection fraction (≥50%) in echocardiography. All patients will undergo body composition analysis and adenosine stress echocardiography with the evaluation of coronary artery blood flow by Doppler echocardiography and maximal oxygen consumption (VO2 max) by cardiopulmonary exercise test (CPET). Left ventricular end-diastolic pressure will be assessed during coronary angiography. Coronary flow reserve (CFR) is defined as the ratio of peak to baseline mean diastolic velocity of coronary blood flow. The correlation of CFR and body composition with cardiopulmonary exercise capacity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80
* Typical/atypical chest pain or ischemic symptoms including dyspnea
* No significant coronary artery stenosis (>50% stenosis) in coronary angiography or computed tomography
* Left ventricular ejection fraction ≥50%

Exclusion Criteria:

* More than moderate valvular heart disease
* Congenital heart disease
* Chronic renal failure (estimated glomerular filtration rate <30 ml/min/1.73m2) or end-stage renal failure undergoing hemodialysis or peritoneal dialysis
* Asthma, chronic obstructive pulmonary disease and primary pulmonary hypertension
* Receiving anticancer drugs
* Vasculitis associated with autoimmune diseases
* Patients with difficulty in performing exercise load evaluation (treadmill, bicycle ergometer)
* Atrial fibrillation
* Atrioventricular block with more than second degrees, symptomatic bradycardia, cryo-node failure syndrome, Wolff-Parkinson-White (WPW) patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of coronary blood flow with cardiopulmonary exercise capacity | up to day 14
  Coronary blood flow is assessed by coronary flow reserve (CFR), which is defined as peak to baseline mean diastolic velocity of coronary flow.
  In regard to cardiopulmonary exercise capacity, maximal oxygen consumption (VO2max) will be assessed.
Correlation of body composition with cardiopulmonary exercise capacity | up to day 14
  In body composition analysis, skeletal muscle mass and body fat mass will be assessed.
  In regard to cardiopulmonary exercise capacity, maximal oxygen consumption (VO2max) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SR, Cho DH, Kim MN, Park SM. Rationale and Study Design of Differences in Cardiopulmonary Exercise Capacity According to Coronary Microvascular Dysfunction and Body Composition in Patients with Suspected Heart Failure with Preserved Ejection Fraction. Int J Heart Fail. 2021 Sep 14;3(4):237-243. doi: 10.36628/ijhf.2021.0029. eCollection 2021 Oct. PMID 36262558